CLINICAL TRIAL: NCT04961606
Title: Qualitative Research on the Influencing Factors of Exercise Adherence of Home-based Cardiac Rehabilitation in Patients With Coronary Artery Disease
Brief Title: Exercise Adherence of Home-based Cardiac Rehabilitation
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2020452
Record Dates: First submitted 2021-06-27; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Home-based cardiac rehabilitation; Exercise adherence
MeSH Terms: conditions — Coronary Artery Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with coronary artery disease
  Interventions: Other: interview
- medical professionals
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — semi-structured individual interview

SUMMARY:
The study explored the influencing factors of exercise adherence of home-based cardiac rehabilitation in patients with coronary artery disease.

DETAILED DESCRIPTION:
The study used a qualitative exploratory design. Informants were recruited by purposive sampling. Semi-structured individual interviews were conducted among patients with coronary artery disease and medical professionals in home-based cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of coronary artery disease;
* Age ≤75 years old;
* Participated in home-based cardiac rehabilitation ≥12 weeks;
* Have good language skills;
* Volunteer to participate in this study.

Exclusion Criteria:

* Have other serious acute or chronic diseases;
* A previous history of mental illness or a positive family history of mental illness;
* Have severe audio-visual or speech impairments that may affect understanding and answering questions.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with coronary artery disease and medical professionals in home-based cardiac rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Influencing factors of exercise adherence | The influencing factors of exercise adherence in home-based cardiac rehabilitation will be measured by the construct of the theory of planned behavior through study completion, an average of 5 months
  Influencing factors of exercise adherence in home-based cardiac rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No